CLINICAL TRIAL: NCT00740740
Title: Biological and Biochemical Markers of Aneurysm Wall Degradation; Towards Non-Invasive Wall Strength Analysis.
Brief Title: Biomarkers of Aneurysm Wall Strength
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Radboud University Nijmegen Medical Centre (M. Truijers MD), Radboud University Nijmegen Medical Centre
Other Study IDs: Wallstrength_01
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2008-08-25 (Estimated); Status verified 2008-08

CONDITIONS: Abdominal Aortic Aneurysm
Keywords: Aneurysm; Rupture
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Aneurysm; Rupture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, urine, tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Patients scheduled for elective conventional aneurysm repair
- 2: Patients scheduled for emergent conventional aneurysm repair
- 3: Patients scheduled for aortic bypass surgery

SUMMARY:
The purpose of this study is to identify possible in vivo biochemical and biological markers related to aortic wall strength.

DETAILED DESCRIPTION:
Rupture of an Abdominal Aortic Aneurysm (AAA) is potentially lethal. prophylactic surgical repair is therefore warranted when the risk of rupture exceeds the risk of complications following surgery. Aneurysm rupture occurs when the forces (stress) acting on the aneurysm wall surpass aneurysm wall strength. Information on both wall stress and strength might therefore improve rupture risk assessment and patient selection for prophylactic repair. Although aneurysm wall stress calculations are possible, no in vivo method exists to determine aneurysm wall strength. This study was designed to identify possible biomarkers of aneurysm wall strength

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for transabdominal aortic surgery

Exclusion Criteria:

* Patient characteristics and aneurysm anatomy suitable for endovascular repair
* Previous aortic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary care clinic. Patients scheduled for transbadominal aortic surgery
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Aneurysm wall strength | Post-operative

SECONDARY OUTCOMES:
Extra Cellular Matrix components (Glucoaminoglycans) | post-operative
Biochemical blood analysis | post-operative
MMP content | post-operative
Degree of inflammation | Post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Jan Blankensteijn, Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Alysis Zorggroep, Rijnstate Hospital, Arnhem, Gelderland
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland